CLINICAL TRIAL: NCT00478634
Title: An Open-label, Multicenter Phase 1 Study Investigating the Combination of RAD001, Cetuximab and Irinotecan as Second-line Therapy After FOLFOX (or XELOX) Plus Bevacizumab (if Given as Part of Local Standard Practice) in Patient With Metastatic Colorectal Adenocarcinoma
Brief Title: A Phase 1 Study Investigating the Combination of RAD001, Cetuximab and Irinotecan as Second-line Therapy After FOLFOX (or XELOX) Plus Bevacizumab in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2242
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
Keywords: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumors; Neoplasms, Colorectal
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Everolimus; Cetuximab; Irinotecan

ARMS (2):
- A1: RAD001 + cetuximab + irinotecan (Experimental): RAD001 30mg weekly oral, 400mg/m2, loading i.v. (250mg/m2 for subsequent weekly dose i.v.), 350mg/m2 every 3 weeks i.v.
  Interventions: Drug: RAD001, Cetuximab, Irinotecan
- B1 dose: RAD001 + cetuximab + irinotecan (Experimental): RAD001 30mg weekly oral, 400mg/m2 loading i.v (250mg/m2 for subsequent weekly dose i.v.), 250mg/m2 every 3 weeks i.v.
  Interventions: Drug: RAD001, Cetuximab, Irinotecan

INTERVENTIONS:
Drug: RAD001, Cetuximab, Irinotecan

SUMMARY:
This study will assess the safety of RAD001 when given together with cetuximab and irinotecan

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years old and ≤ 65 years old.
* Patients with metastatic CRC. Confirmation of CRC diagnosis by histological or cytological specimen from original resection of primary tumor.
* Patients who progressed despite prior therapy with FOLFOX (5FU and oxaliplatin) plus bevacizumab or XELOX (capecitabine and oxaliplatin) plus bevacizumab.
* Patients with at least one measurable lesion by RECIST as determined by Computer Tomography (CT) Scan, Magnetic Resonance Imaging (MRI) or physical examination.
* Patients with a WHO performance status of 0 or 1.

Exclusion criteria:

* Patients with Gilbert's syndrome or any other syndrome associated with deficient glucoronidation of bilirubin.
* Patients who are homozygous for the UGT1A1*28 allele as determined by sequencing.
* Patients who have received previous irinotecan-based therapy.
* Prior treatment with an mTOR inhibitor.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | at end of cycle 2
  each cycle was 21 days

SECONDARY OUTCOMES:
Pharmacokinetics of RAD001, Irinotecan and SN-38
Progressions Free Survival
Overall Survival
Objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- United States (16):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Comprehensive nBlood and Cancer Care, Bakersfield, California
  - UCSD - Moores Cancer Center, La Jolla, California
  - Comprehensive Cancer Care, Los Angeles, California
  - North Valley Hematology/Oncology Medical Group: The Thomas & Dorothy Leavey Cancer Center, Northridge, California
  - Cancer Care Associates Medical Group, Inc., Redondo Beach, California
  - Norwalk Hospital, Norwalk, Connecticut
  - Gerogetown University Lombardi Cancer Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Oncology Specialists, Park Ridge, Illinois
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Richmond University Medical Center, Staten Island, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Oncology/Hematology Associates, Bethlehem, Pennsylvania
  - Arlington Cancer Center, Arlington, Texas